CLINICAL TRIAL: NCT04119128
Title: Effects of Transcranial Direct Current Stimulation (tDCS) on Fatigue in Patients With Primary Sjogren's Syndrome: a Double-blinded Randomized Trial
Brief Title: tDCS for Fatigue in Sjogren's Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: University of Pittsburgh (Other); Universidade Federal do Amapá (Other)
Responsible Party: Principal Investigator, Ana Carolina Pereira Nunes Pinto, MSc, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FederalUnivOfSaoPaulo
Record Dates: First submitted 2019-10-04; First posted 2019-10-08 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Sjogren's Syndrome
Keywords: Sjogren's Syndrome; fatigue; tDCS
MeSH Terms: conditions — Sjogren's Syndrome; Fatigue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Active Comparator): Patients in this group will receive 5 active sessions of low-intensity transcranial electrical stimulation for 20 minutes.
  Interventions: Device: Active Transcranial Direct Current Stimulation
- Sham tDCS (Sham Comparator): Patients in this group will receive 5 sessions of sham transcranial electrical stimulation for 20 minutes.
  Interventions: Device: Sham Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Active Transcranial Direct Current Stimulation — Subjects will undergo 5 sessions of tDCS of up to 2mA, at 20 minutes per session, 1x per day. During active stimulation, the current will be active for the full 20 minutes.
  Arms: Active tDCS
Device: Sham Transcranial Direct Current Stimulation — Subjects will undergo 5 sessions of tDCS, at 20 minutes per session, 1x per day. For sham tDCS, electrodes will be placed the same way as in the intervention group, for 20 minutes. However, the stimulator will deliver 2mA of current for only 30s. The current will not be active for the rest of the 20 minutes.
  Arms: Sham tDCS

SUMMARY:
Sjogren's Syndrome (SS) is an autoimune disease of unknown etiology characterized by lymphocytic infiltration of the exocrine glands and other organs. patients usually presents with xerophthalmia, xerostomia, fatigue and other symptoms. Fatigue has often been reported as the biggest problem and the most difficult symptom patients have to deal with. Fatigue management in pSS is difficult. However, in other diseases such as Parkinson disease, post-polio syndrome and multiple sclerosis the use of Transcranial Direct Current Stimulation (tDCS) has recently been studied and has shown effectiveness. The overarching objective of this study is to examine the effect of a tDCS protocol in patients with pSS.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Age between 18 and 65 years old;
* Diagnosis of primary Sjogren's Syndrome according to American-European Criteria;
* Stable pharmacological therapy for at least 3 months;
* Complaints of fatigue as assessed by Fatigue Severity Scale (FSS>5).
* Complaints of fatigue for more than 3 months.

Exclusion Criteria:

* Heart, coronary, respiratory, renal, or hepatic uncompensated insufficiencies;
* Uncompensated systemic arterial hypertension;
* Unable to answer the questionnaires.
* Severe depression (with a score > 30 in the Beck Depression Inventory)
* History of epilepsy or syncope
* Implanted brain metallic devices
* Established cognitive impairment
* Traumatic brain injury with residual neurological deficits

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Change in Fatigue | Change in fatigue from baseline to 15 days after the end of stimulation.
  Will be assessed with Fatigue Severity Scale (FSS). FSS is a 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle in patients with a variety of disorders. The items are scored on a 7-point scale. Higher values indicate higher severity of fatigue.

SECONDARY OUTCOMES:
Change in Profile of Fatigue | Will be measured at baseline, on the 5th day of stimulation (immediately after the end of stimulation), 15 days after the end of stimulation and 30 days after the end of stimulation
  Will be assessed with Profile of Fatigue and Discomfort - Sicca Symptoms Inventory (short form) (Profad-SSI-SF). Profad-SSI-SF is a 19-item questionnaire assessing the subjective aspects of the symptoms of Sjogren's Syndrome, including fatigue, based on the patient's perception. The items are scored from 0 to 7 points. Higher values indicate higher severity of fatigue.
Change in Symptoms severity | Will be measured at baseline, on the 5th day of stimulation (immediately after the end of stimulation), 15 days after the end of stimulation and 30 days after the end of stimulation
  Will be assessed with EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI). ESSPRI is a very simple index designed to measure patients' symptoms of patients with Sjogren's Syndrome. ESSPRI is completed by the patient and it contains just three items to be given a score between 0-10: for pain, fatigue and dryness, the final ESSPRI score is the mean of all three scores and therefore also between 0-10. Higher values indicate higher severity of symptoms.
Change in Quality of Life | Will be measured at baseline, on the 5th day of stimulation (immediately after the end of stimulation), 15 days after the end of stimulation and 30 days after the end of stimulation
  Will be assessed with 12-Item Short-Form (SF-12). The SF-12 is a multipurpose short form survey with 12 questions. The SF-12 is weighted and summed to provide easily interpretable scales for physical and mental health. Physical and Mental Health Composite Scores (PCS & MCS) are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Change in Patient Global Assessment | Will be measured after the 1st, 5th day of stimulation, 15 days after the end of stimulation and 30 days after the end of stimulation.
  Subjects will rate their global assessment using verbal response and a visual analog scale (0-10). They will rate: Global health.
Change in Adverse Events | Will be measured up to 30 days after the end of stimulation.
  Subjects will complete a structured questionnaire to assess potential adverse events of stimulation

OTHER OUTCOMES:
Change in Hypothalamic-pituitary-adrenal (HPA) axis activity | Will be measured immediately before and immediately after the first day of stimulation and immediately before and immediately after the last day (5th) day of stimulation.
  Salivary cortisol
Change in Sleep Quality | Will be measured at baseline, on the 5th day of stimulation (immediately after the end of stimulation), 15 days after the end of stimulation and 30 days after the end of stimulation
  Will be assessed with Pittsburgh Sleep Quality Index (PSQI). PSQI is a self-report questionnaire that assesses sleep quality. It's composed by nineteen individual items that generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score. The global PSQI score ranges from 0 to 21, where lower scores denote a healthier sleep quality.
Change in Depression | Will be measured at baseline, on the 5th day of stimulation (immediately after the end of stimulation), 15 days after the end of stimulation and 30 days after the end of stimulation
  Will be assessed using Beck Depression Inventory (BDI). BDI is a 21-item self-report inventory, for measuring the severity of depression. The items are scored from 0 to 3 points. Higher values indicate higher severity of depression.
Change in Patient Self Assessment | Will be measured at baseline, on the 5th day of stimulation (immediately after the end of stimulation), 15 days after the end of stimulation and 30 days after the end of stimulation
  Subjects will rate their assessment using verbal response and a visual analog scale (0-10). They will rate: Anxiety, stress and sleepiness.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Pinto, MSc, Principal Investigator — Federal University of Amapa/Federal University of Sao Paulo
Locations (1):
- FUSaoPaulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all outcomes will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available after 6 months of study completion.
Access Criteria: Data access request will be analysed and requestors will be required to sign a Data Access Agreement